CLINICAL TRIAL: NCT00408135
Title: Evaluation of the Safety, Efficacy and Acceptability of HMR 3647 (20％ Fine Granules 1 g Sachet) in Children With Infections
Brief Title: Japanese Study Evaluating Safety, Efficacy and Acceptability of Telithromycin in Children With Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFC6371; HMR3647B/3104
Record Dates: First submitted 2006-12-05; First posted 2006-12-06 (Estimated); Last update posted 2009-04-03 (Estimated); Status verified 2009-04

CONDITIONS: Infections; Child
Keywords: Respiratory Tract Infections; Skin Diseases; Sinusitis
MeSH Terms: conditions — Infections; Respiratory Tract Infections; Skin Diseases; Sinusitis | interventions — telithromycin

INTERVENTIONS:
Drug: telithromycin (HMR3647)

SUMMARY:
The primary objective is to assess the safety of telithromycin (HMR 3647) (20% fine granules) 1g filling sachet in children with infections (Respiratory tract infections, Dermatological infections, Otorhinolaryngological infections, Dentistry/Oral surgery infections).

Secondary objectives are to assess the clinical efficacy, bacteriological efficacy and acceptability of telithromycin (20% fine granules) 1g filling sachet in children with infections.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients of weight from 7.0 kg.
* For respiratory tract infections:subjects diagnosed with mild or moderate respiratory tract infection (excluding pneumonia) based on a fever (≥ 38°C) or C-Reactive Protein positive, clinical symptoms/signs, and laboratory findings.
* For dermatological infections: subjects diagnosed with mild or moderate dermatological infection in terms of clinical symptoms/signs and laboratory findings.
* For otorhinolaryngological infections:subjects with purulent / mucopurulent rhinorrhea and postrhinorrhea, subjects diagnosed with mild or moderate otorhinolaryngological infection in terms of clinical symptoms/signs and laboratory findings
* For dental / oral surgical infections: subjects who have formed obstructive abscess and diagnosed with mild or moderate dental / oral surgical infection

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 111 (Actual)
Dates: Start 2004-08; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Safety evaluation: presence/absence of subjective/objective symptoms and abnormal laboratory findings (abnormal changes of parameters in general hematological tests and blood biochemical tests).

SECONDARY OUTCOMES:
Clinical efficacy:change in the symptoms and signs at end of therapy visit and at the test of cure visit

CONTACTS AND LOCATIONS:
Overall Officials: Norifumi Yamamoto, Study Director — sanofi-aventis Japan
Locations (1):
- Sanofi-Aventis, Tokyo, Japan